CLINICAL TRIAL: NCT07318948
Title: BALANCE Trial Protocol - Blood Pressure Lowering and Thrombolysis: Concurrent vs Sequential Management in Acute Ischemic Stroke
Brief Title: BALANCE Trial Domain Within the ACT-GLOBAL Adaptive Platform Trial-NCT06352632
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bo Wu (Other)
Collaborators: West China Hospital (Other); Mianyang Central Hospital (Other); Panzhihua Central Hospital (Other); The First People's Hospital of Ziyang (Unknown); Zigong The Fourth People's Hospital (Other); Zigong No.1 Peoples Hospital (Other)
Responsible Party: Sponsor-Investigator, Bo Wu, Dr., West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025(No.2280)
Record Dates: First submitted 2025-12-08; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Thrombolysis; Blood Management
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Different sequences of blood pressure management and intravenous thrombolysis.
Who Masked: Outcomes Assessor
Masking Description: The neurologists and radiologists at the central imaging core laboratory who are responsible for adjudicating all imaging endpoints, including symptomatic intracerebral hemorrhage (sICH).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sequential Arm (No Intervention): 1. Antihypertensive Therapy: Immediately after randomization, intravenous antihypertensive therapy is initiated to actively lower the patient's blood pressure to below the guideline recommended range.
  2. Thrombolysis: Once the blood pressure is confirmed to be at or below the guideline recommended range, intravenous thrombolysis (alteplase or tenecteplase, per local standard of care) is administered.
- Conccurent Arm (Experimental): 1. Thrombolysis: Immediately after randomization, intravenous thrombolysis (alteplase or tenecteplase, per local standard of care) is administered as per local practice.
  2. Antihypertensive Therapy: As soon as feasible after the start of thrombolysis, intravenous antihypertensive therapy is initiated with the goal of lowering blood pressure to below guideline recommended range. (e.g. China: 180/100 mmHg; U.S./Canada/Europe: 185/110 mmHg).
  Interventions: Other: Concurrent Thrombolysis

INTERVENTIONS:
Other: Concurrent Thrombolysis — Lowering the blood pressure and undergoing thrombolysis at the same time while the partipants blood pressure is higher than 185/110 mmHg or 180/100 mmHg.
  Arms: Conccurent Arm

SUMMARY:
Elevated blood pressure (BP) is nearly universal in acute ischemic stroke (AIS) and critically influences eligibility for intravenous thrombolysis; however, current guidelines-requiring BP reduction to below 185/110 mmHg before treatment-lack robust evidence and may delay reperfusion in a time-sensitive therapy, potentially worsening outcomes. Emerging data suggest that aggressive pre-thrombolysis BP lowering does not reduce hemorrhage risk and might impair recovery, highlighting the need to avoid large BP fluctuations. Yet it remains uncertain whether initiating thrombolysis concurrently with antihypertensive therapy is safer and more effective than the standard sequential approach, particularly in patients with markedly elevated but not extreme BP (systolic <220 mmHg).

To address this gap, the BALANCE trial is a prospective, multicenter, randomized controlled study enrolling AIS patients within 4.5 hours of onset whose pre-thrombolysis BP exceeds regional guideline thresholds (e.g., >180/100 mmHg in China or >185/110 mmHg internationally) but is <220 mmHg and who are otherwise eligible for thrombolysis. Patients are randomized to either: (1) concurrent management-immediate thrombolysis with simultaneous IV antihypertensive therapy to gradually lower BP-or (2) sequential management-antihypertensive treatment first, followed by thrombolysis only after BP reaches target. The primary endpoint is a hierarchical composite analyzed using the win ratio, prioritizing: (1) functional outcome (90-day mRS distribution), (2) major safety (symptomatic intracerebral hemorrhage within 7 days per SITS-MOST criteria), and (3) process efficiency (door-to-needle time).

Conducted across 80-100 global stroke centers, BALANCE aims to provide definitive evidence to optimize BP management and improve outcomes in AIS patients with elevated BP.

DETAILED DESCRIPTION:
Hypertension is the most common physiological abnormality in patients presenting with acute ischemic stroke (AIS), and elevated blood pressure (BP) plays a critical role in determining eligibility and timing for intravenous thrombolysis.

Current international guidelines recommend lowering BP to below 185/110 mmHg before administering thrombolytic therapy, a process that requires antihypertensive treatment and inevitably delays thrombolysis. However, this recommendation lacks robust evidence. Meanwhile, because the effectiveness of thrombolysis is highly time-dependent, these BP-lowering delays may worsen clinical outcomes by prolonging door-to-needle time and delaying reperfusion.

On the other hand, recent prospective studies on blood pressure management before and after thrombolysis and thrombectomy have shown that lower BP levels do not significantly reduce the risk of hemorrhage and may lead to poorer long-term outcomes. Although these studies compared BP ranges below 180 or 185 mmHg, it remains unclear whether this pattern applies to patients with severely elevated BP. These findings suggest the importance of avoiding large and rapid BP fluctuations. Initiating thrombolysis after BP reduction could result in significant BP fluctuations and prolonged periods of low BP post-thrombolysis.

Given the lack of high-quality evidence on optimal treatment strategies for patients with pre-thrombolysis hypertension, an alternative concurrent BP management strategy has been proposed. This approach involves initiating thrombolysis and antihypertensive treatment simultaneously. By doing so, it aims to minimize treatment delays while maintaining BP control within accepted post-thrombolysis targets. However, concerns exist about whether initiating thrombolysis at higher-than-recommended BP levels increases the risk of symptomatic intracerebral hemorrhage or other complications. Consequently, substantial clinical uncertainty exists regarding which strategy-concurrent or sequential BP management-is superior for patients.

The BALANCE trial is a prospective, multicenter, randomized controlled study compare the effectiveness and safety between concurrent and sequential strategies. The concurrent strategy involves immediate initiation of intravenous thrombolysis, accompanied by simultaneous IV antihypertensive therapy to gradually lower BP during and after thrombolysis. In contrast, the sequential strategy starts with antihypertensive treatment, and thrombolysis is withheld until BP falls within guideline-recommended limits. AIS patients presenting within 4.5 hours of symptom onset with pre-thrombolysis BP exceeding guideline-recommended ranges (e.g., China: 180/100 mmHg; U.S./Canada/Europe: 185/110 mmHg) but below 220 mmHg, and who are otherwise eligible for intravenous thrombolysis, will be enrolled across 80-100 stroke centers worldwide. The primary endpoint is a hierarchical composite outcome analyzed using the win ratio method. It comprises three components, prioritized in the following order: (1) functional outcome, defined as the distribution of modified Rankin Scale (mRS) scores at 90 days after randomization; (2) major safety, defined as the occurrence of symptomatic intracerebral hemorrhage (sICH) within 7 days after randomization according to the SITS-MOST criteria; and (3) process efficiency, defined as door-to-needle time (DNT)-the interval from emergency department arrival to the start of thrombolytic infusion. In pairwise comparisons between treatment groups, a patient "wins" if they have a better outcome on the highest-priority component where a difference exists.

By evaluating these two fundamentally different management pathways, the BALANCE trial seeks to generate definitive evidence that may inform future guideline recommendations and optimize care for patients with acute ischemic stroke and elevated blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Clinical diagnosis of acute ischemic stroke with a clearly defined time of symptom onset or last known well, allowing for randomization within 4.5 hours.
* The treating physician has made the decision to treat the patient with intravenous thrombolysis.
* Elevated blood pressure, defined as: Pre-thrombolysis BP exceeds guideline-recommended range (e.g. China: 180/100 mmHg; U.S./Canada/Europe: 185/110 mmHg), but below 220 mmHg.

  *The qualifying blood pressure must be confirmed by two separate measurements taken at least one minute apart from the same arm, using an appropriately sized cuff while the patient is in a supine or semi-recumbent position.
* Informed consent is obtained from the patient or a legally authorized representative in accordance with local regulations. A deferred or waiver of consent model will be used where permitted by local ethics committees for emergency research.

Exclusion Criteria:

* Any condition that, in the judgment of the investigator, would preclude follow-up or interfere with outcome assessment (e.g., end-stage malignancy, severe multi-organ failure).
* The patient is pregnant or breastfeeding.
* Concurrent enrollment in another interventional trial where the intervention is likely to confound the study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint: A Justification for the Hierarchical Win Ratio | 90-day
  The win ratio is a patient-centered statistical method that allows for the comparison of treatment arms across several prioritized outcomes. It provides a more holistic assessment of the net clinical benefit. The hierarchy is ordered based on clinical importance:
  1. Functional Outcome: Defined as the distribution in scores on the modified Rankin scale (mRS) at 90 days after randomization.
  2. Major Safety: Defined as the sICH occurrence within 7 days after randomization, based on SITS-MOST criteria.
  Process Efficiency: Defined as the time between emergency department entry to thrombolysis start (DNT).

SECONDARY OUTCOMES:
Excellent Functional Outcome | 90-day
  The proportion of patients with an mRS score of 0-1 at 90 days.
Good Functional Outcome | 90-day
  The proportion of patients with an mRS score of 0-2 at 90 days.
Distribution of Functional Outcome | 90-day
  The mRS score at 90 days and the utility weighted mRS.
Quality of Life at 90 days | 90-day
  Quality of Life measured using the EQ-5D-5L at 90 days.
Neurological Status at 72 Hours | 72±12 hours
  The National Institutes of Health Stroke Scale (NIHSS) score assessed between 72±12 hours post-randomization.
Early Neurological Improvement | 72±12 hour
  Defined as achieving an NIHSS score of 0-1 or a decrease of ≥4 points from the baseline NIHSS score at the 72±12 hour assessment.
Mortality | 90-day
  All-cause mortality at 90 days.
Malignant Cerebral Edema | 90-day
  The incidence of malignant edema, adjudicated by the central imaging core lab according to follow-up imaging and medical history.
Process Metrics | 24-hour
  DNT, the time between emergency department entry to thrombolysis start.

OTHER OUTCOMES:
sICH occurrence | 7-day
  The primary definition of sICH is based on SITS-MOST criteria. sICH will be diagnosed only when both radiological and clinical criteria are met:
  Radiological criterion: Presence of parenchymal hematoma type 2 (PH2) on follow-up neuroimaging, defined as a dense hematoma.
  Clinical criterion: Neurological deterioration of ≥4 points on the NIH Stroke Scale (NIHSS) compared with baseline, or death.
  The sensitivity analysis for sICH will use the NINDS definition. sICH will be diagnosed only when both radiological and clinical criteria are met: Radiological criterion: Any intracranial hemorrhage (including hemorrhagic infarction or parenchymal hematoma). Clinical criterion: Any worsening of neurological status, with no minimum NIHSS threshold specified.
Any Intracerebral Hemorrhage | 7-day
  Any evidence of ICH on follow-up imaging up to 7 days.
Hemorrhagic Event Classification | 7-day
  All follow-up imaging will be systematically assessed by the central core lab using the Heidelberg Bleeding Classification to categorize any hemorrhagic event.
Early Mortality | 7-day
  All-cause mortality at 7 days and in-hospital mortality.
Serious Adverse Events (SAEs) | From randomization through Day 4 or hospital discharge, whichever occurs first.
  In line with the pragmatic design of the trial, the formal collection and reporting of SAEs will be limited to the period from randomization through Day 4 or hospital discharge, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Bijoy Menon, MD, Phd, Principal Investigator — University of Calgary; Bo Wu, MD, PhD, Principal Investigator — West China Hospital
Locations (1):
- Bo Wu, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
This study will include individual information from multicenter and multination. To protect the participants' privacy and follow the guidelines of other center or nations' ethical committee, we don't provide or share IPD with other reasearchers.